CLINICAL TRIAL: NCT00605826
Title: A Randomized, Subject and Evaluator Blinded, Sham Controlled, Multicenter Study to Evaluate Efficacy and Safety of NASHA/Dx for the Treatment of Fecal Incontinence
Brief Title: A Randomized, Blinded, Multicenter Study to Evaluate NASHA/Dx for the Treatment of Fecal Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Collaborators: Oceana Therapeutics, Inc. (Industry); Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 33DA0404
Record Dates: First submitted 2008-01-09; First posted 2008-01-31 (Estimated); Results first posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Blinded injection of NASHA/Dx gel at randomization. (Experimental): Blinded injection of NASHA/Dx (Solesta) Gel. For each treatment, a series of 4 equally spaced injections with 1 mL of Solesta into the anal canal. Subjects will be followed for 6 months during the blinded phase. During a subsequent open phase, these subjects will be followed to Month 36 (ie, for an additional 30 months).
  Interventions: Device: NASHA/Dx (Solesta) Gel
- Blinded sham inject. at randomization (Sham Comparator): Blinded sham injection (needle stick with empty syringes). For each treatment, a series of 4 equally spaced Sham injections (needle sticks) into the anal canal. Subjects will be followed for 6 months during the blinded phase.
  Sham-treated subjects have the option to receive open-label injection of NASHA/Dx (Solesta) Gel at the 6-month time point following completion of the blinded phase (ie, blinded sham injection at randomization + NASHA/Dx Gel at 6 months). Following injection of NASHA/Dx gel at the start of the open phase, these subjects will be followed to Month 30 (ie, for an additional 24 months).
  Interventions: Device: Sham Injection
- Blinded Sham Inject. at Randomization + NASHA/Dx Gel at 6 mo. (Other): Blinded sham injection at randomization. Subjects will be followed for 6 months during the blinded phase.
  Sham-treated subjects have the option to receive open-label injection of NASHA/Dx (Solesta) Gel at the 6-month time point following completion of the blinded phase (ie, blinded sham injection at randomization + NASHA/Dx Gel at 6 months). Following injection of NASHA/Dx gel at the start of the open phase, these subjects will be followed to Month 30 (ie, for an additional 24 months).
  Interventions: Device: NASHA/Dx (Solesta) Gel; Device: Sham Injection

INTERVENTIONS:
Device: NASHA/Dx (Solesta) Gel — Injection of 4 x 1ml of NASHA/Dx Gel at the start of the blinded phase.
  Other Names: Solesta
  Arms: Blinded Sham Inject. at Randomization + NASHA/Dx Gel at 6 mo.; Blinded injection of NASHA/Dx gel at randomization.
Device: Sham Injection — Sham injection at the start of the blinded phase.
  Arms: Blinded Sham Inject. at Randomization + NASHA/Dx Gel at 6 mo.; Blinded sham inject. at randomization

SUMMARY:
The purpose of this study is to determine the effectiveness and safety of NASHA/Dx when used as an injectable bulking agent in the treatment of fecal incontinence. The study includes a 6-month blinded sham-controlled phase, followed by an open-label phase.

DETAILED DESCRIPTION:
Subjects will be given up to 2 treatments of NASHA/Dx or sham and followed for 6 months from last treatment (ie, one retreatment is permitted at 1 month after the first injection) in the blinded phase of the study. At Month 6, the open phase of the study will begin and subjects on sham will be offered open-label treatment with NASHA/Dx.

Subjects who receive NASHA/Dx at the start of the blinded phase will be followed for up to 36 months from last treatment in the blinded phase. Subjects who receive sham at the start of the blinded phase and then receive open-label NASHA/Dx at Month 6 (start of the open phase) will be followed for another 24 months (equivalent to approximately 30 months from randomization) from last treatment in the open phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age, male or female.
* Screening fecal incontinence severity score (CCFIS).
* Fecal incontinence episodes over a 14-day period.
* Failed conservative treatment for fecal incontinence.

Exclusion Criteria:

* Complete external sphincter disruption.
* Significant anorectal disease.
* Anorectal surgery within the last 12 months prior to the study.
* Active Inflammatory Bowel Disease (IBD).
* Immunodeficiency or receiving immunosuppressive therapy.
* Malignancies in remission for less than 2 years prior to the study.
* Bleeding disorders or receiving anticoagulant therapy.
* Chemotherapy within the last 12 months prior to the study.
* Prior Pelvic radiotherapy.
* Women who are pregnant or breast-feeding, or women of childbearing potential not practicing adequate contraception or planning to stop such contraception within the first year of the study.
* Women within one year post partum.
* Participation in any other clinical study within 3 month prior to the study.
* Hypersensitivity to hyaluronic acid containing products.
* Other severe conditions or in other ways unsuitable to participate according to investigator judgement.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2006-09-07 (Actual); Primary Completion 2009-11-23 (Actual); Study Completion 2009-11-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (8):
  - University of California, San Francisco, Center for Pelvic Physiology, Dept. of Surgery, San Francisco, California
  - University of South Florida College of Medicine, Tampa General Hospital, Tampa, Florida
  - Lahey Clinic, Department of Colon & Rectal Surgery, Burlington, Massachusetts
  - Colon & Rectal Surgery Associates, Minneapolis, Minnesota
  - St. Luke's/Roosevelt Hospital, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Colorectal Surgical Associates, Houston, Texas
  - Salt Lake Research/Center for Colon Rectal Disease, Salt Lake City, Utah
- Chirurgische Klinik Mit Poliklinik, FAU Erlangen-Nurnberg, Erlangen, Germany
- Sweden (3):
  - Kirurgmottagningen Universitetssjukhuset MAS, Malmo
  - Kirurgmottagningen, Danderyds Sjukhus, Stockholm
  - Kirurgkliniken, Uppsala Akademiska Sjukhus, Uppsala
- Castle Hill Hospital, Department of Academic Surgery, Cottingham, East Yorkshire, United Kingdom

REFERENCES:
- [Derived] Graf W, Mellgren A, Matzel KE, Hull T, Johansson C, Bernstein M; NASHA Dx Study Group. Efficacy of dextranomer in stabilised hyaluronic acid for treatment of faecal incontinence: a randomised, sham-controlled trial. Lancet. 2011 Mar 19;377(9770):997-1003. doi: 10.1016/S0140-6736(10)62297-0. PMID 21420555

RESULTS

PARTICIPANT FLOW:
Groups:
- NashaDx/Fecal: NashaDx/Fecal - 4 syringes each containing 1 mL of product
- Sham: Sham - 4 empty syringes
Period: Overall Study
Arm/Group | NashaDx/Fecal | Sham
Started | 136 | 70
Completed | 129 | 60
Not Completed | 7 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NashaDx/Fecal | Sham | Total
Number analyzed (Participants) | 136 | 70 | 206
Age, Continuous [Mean (Full Range); unit: years] | 60.6 [32.8 to 76.0] | 59.2 [29.4 to 75.9] | 60.1 [29.4 to 76.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 61 | 183
  Male | 14 | 9 | 23

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Are Responder50.
Description: Percentage of participants who achieve ≥ 50% reduction in the number of fecal incontinence episodes compared to baseline (Responder50).
Time Frame: 6 months after last blinded treatment
Measure: Count of Participants; unit: Participants
Arm/Group | NashaDx/Fecal | Sham
Number analyzed (Participants) | 136 | 70
Participants | 71 | 21

2. Primary Outcome: Percentage of Participants Who Are Responder25.
Description: Response to treatment at 12 months was defined as a ≥ 25 % reduction in the number of fecal incontinence episodes compared to baseline (Responder25).
Time Frame: 12 months after last treatment
Population: This outcome measure was only analyzed for the NASHA/Dx group.
Measure: Number; unit: percentage of participants
Groups:
- NASHA/Dx Fecal: NASHA/Dx Fecal - 4 syringes each containing 1 mL of product
Arm/Group | NASHA/Dx Fecal
Number analyzed (Participants) | 136
percentage of participants | 69.1

3. Secondary Outcome: Number of Fecal Incontinence Episodes
Description: The number of incontinence episodes collected from a participant incontinence diary spanning a period of 14 days prior to each of the study visits.
Time Frame: up to 6 months after last treatment
Measure: Mean (Standard Error); unit: number of episodes
Arm/Group | NashaDx/Fecal | Sham
Number analyzed (Participants) | 136 | 70
number of episodes | 16.28 (2.15) | 18.53 (5.56)

4. Secondary Outcome: Number of Incontinence Free Days
Description: The number of days with no fecal incontinence episodes (incontinence free days).
Time Frame: up to 6 months after last treatment
Measure: Mean (95% Confidence Interval); unit: incontinence free days
Arm/Group | NashaDx/Fecal | Sham
Number analyzed (Participants) | 136 | 70
incontinence free days | 7.6 [6.68 to 8.52] | 6.48 [5.41 to 7.56]

5. Secondary Outcome: Change From Baseline in Fecal Incontinence Quality of Life Scale (FIQL).
Description: The disease-specific Fecal Incontinence Quality of Life (FIQL) questionnaire is designed to capture the impact of treatment on quality of life for participants suffering from fecal incontinence as it pertains to 4 domains: Lifestyle, Coping/Behavior, Depression/Self perception and Embarrassment. The more the subject is affected by fecal incontinence the lower the value. Hence, a positive change from baseline indicates improvement. Scores range from 1 to 4.
Time Frame: up to 6 months after last treatment
Population: This outcome measure was only analyzed for the NASHA/Dx group.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | NASHA/Dx Fecal
Number analyzed (Participants) | 136
units on a scale
  Lifestyle domain | 0.29 (0.05)
  Coping/Behavior domain | 0.42 (0.05)
  Depression/Self perception domain | 0.30 (0.05)
  Embarrassment domain | 0.45 (0.06)

6. Secondary Outcome: Cleveland Clinic Florida Incontinence Score (CCFIS).
Description: Cleveland Clinic Florida Incontinence Score (CCFIS) score was based on a participant interview using standardized questions regarding incidence and type of incontinence (solid, liquid or gas), pad usage and lifestyle alterations during the past month. The score ranged from 0 (perfect) to 20 (complete incontinence)
Time Frame: up to 6 months after last treatment
Population: This outcome measure was only analyzed for the NASHA/Dx group.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | NASHA/Dx Fecal
Number analyzed (Participants) | 136
units on a scale | -2.45 (0.31)

ADVERSE EVENTS:
Time Frame: 36 months
Description: Adverse events were assessed in all treated subjects and not by treatment group.
Groups:
- Overall: Adverse events were assessed overall and not by randomized treatment group
Arm/Group | Overall
Serious Adverse Events (participants affected / at risk) | 31/206
Other Adverse Events (participants affected / at risk) | 78/206
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall (N=206)
Abdominal pain (Gastrointestinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Arterial senosis limb (Vascular disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Atrial fibrillation (Cardiac disorders) | 1
Back pain (General disorders) | 2
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carotid artery stenosis (Vascular disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Chest pain (General disorders) | 2
Cholelithiasis (Gastrointestinal disorders) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Enterocele (General disorders) | 1
Gastroenteritis (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2
Multiple endocrine adenomatosis Type II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Nausea (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1
Rectal prolapse (Gastrointestinal disorders) | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal abscess (Gastrointestinal disorders) | 2
E. coli bacteremia (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Overall (N=206)
Injection site haemorrhage (General disorders) | 16
Proctalgia (Gastrointestinal disorders) | 33
Rectal haemorrhage (Gastrointestinal disorders) | 15
Pyrexia (General disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.